CLINICAL TRIAL: NCT00620373
Title: Evaluation of Low-dose Molecular Breast Imaging as a Screening Tool in Women With Mammographically Dense Breasts and Increased Risk of Breast Cancer
Brief Title: Molecular Breast Imaging as a Screening Tool for Women With Dense Breasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Deborah Rhodes, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1337-05 Part A; Susan G. Komen Foundation
Record Dates: First submitted 2007-12-21; First posted 2008-02-21 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: Dense breast tissue; Breast Cancer Screening; Molecular Breast Imaging; Breast Cancer; Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mammography and Molecular Breast Imaging (Experimental): Participants underwent conventional mammography and molecular breast imaging after a 740-millibecquerel (mBQ) (20-mCi) Technetium (99mTc) sestamibi injection.
  Interventions: Device: Molecular Breast Imaging; Device: Conventional Mammography; Drug: Technetium (99mTc) sestamibi

INTERVENTIONS:
Device: Molecular Breast Imaging — Molecular breast imaging is a new nuclear medicine technique for imaging the breast. It uses small field of view semiconductor-based gamma cameras that use Cadmium Zinc Telluride detectors. These have superior spatial and energy resolution to conventional sodium iodide detectors.
Device: Conventional Mammography — Mammography is the process of using low-energy X-rays (usually around 30 kVp) to examine the human breast and is used as a diagnostic and a screening tool.
Drug: Technetium (99mTc) sestamibi — Technetium (99mTc) sestamibi is a pharmaceutical agent used in nuclear medicine imaging. The drug is a coordination complex consisting of the radioisotope technetium-99m bound to six methoxyisobutylisonitrile (MIBI) ligands.
  Other Names: Cardiolite

SUMMARY:
We aim to compare the sensitivity of mammography to the sensitivity of Molecular Breast Imaging (a new gamma-camera based breast imaging technology) in women with dense breast tissue who are at increased risk for breast cancer.

DETAILED DESCRIPTION:
The sensitivity of conventional mammography (MMO) is poor in women with mammographically dense breast parenchyma. We have developed Molecular Breast Imaging (MBI) - a new technique which utilizes a Cadmium-Zinc-Telluride (CZT) gamma camera for scintimammography that has a high sensitivity (~90%) for the detection of breast cancers independent of breast density.

The aim of this study is to demonstrate the utility of MBI as an adjunct screening modality for the detection of occult breast cancers in women with mammographically dense breast tissue. Initial recruitment will be from the pool of patients awaiting a screening mammogram in the Department of Radiology at Mayo Clinic Rochester. All patients will have a screening MMO and an MBI study. Patients with positive studies (MBI or MMO) will undergo additional diagnostic studies. At 15 months post-recruitment, all patients will be contacted by phone or mail to determine whether subsequent to their study, there has been any change in their breast status.

ELIGIBILITY:
Inclusion Criteria:

1. Past prior screening mammography (SM) interpreted as negative or benign (This screening must have been performed at Mayo Clinic Rochester, Minnesota).
2. Past prior SM interpreted as heterogeneously dense or extremely dense (This screening must have been performed at Mayo Clinic Rochester, Minnesota).
3. Women younger than 50 years who had not undergone prior mammography, as most of these women have dense breasts.
4. Subjects had to have at least one of the following risk factors:

   1. Known mutation in breast cancer susceptibility gene 1 (BRCA1) or breast cancer susceptibility gene 2 (BRCA2)
   2. History of chest, mediastinal, or axillary irradiation
   3. Personal history of breast cancer
   4. History of prior biopsy showing atypical ductal hyperplasia, atypical lobular hyperplasia, lobular carcinoma in situ, or atypical papilloma
   5. Gail or Claus model lifetime risk greater than or equal to 20%
   6. Gail model 5 year risk greater or equal to 2.5%
   7. Gail model 5 year risk greater or equal to 1.6%
   8. One first-degree relative with history of breast cancer
   9. Two second-degree relatives with history of breast cancer

Exclusion Criteria:

1. They are unable to understand and sign the consent form
2. They are pregnant or lactating
3. They are physically unable to sit upright and still for 40 minutes.
4. They have self-reported signs or symptoms of breast cancer (palpable mass, bloody nipple discharge, axillary mass etc.).
5. They have had needle biopsy within 3 months, or breast surgery within 1 year prior to the study.
6. They are currently taking tamoxifen, evista (raloxifene), or an aromatase inhibitor for adjuvant therapy or chemoprevention.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 969 (Actual)
Dates: Start 2005-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Rhodes, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Rhodes DJ, Hruska CB, Phillips SW, Whaley DH, O'Connor MK. Dedicated dual-head gamma imaging for breast cancer screening in women with mammographically dense breasts. Radiology. 2011 Jan;258(1):106-18. doi: 10.1148/radiol.10100625. Epub 2010 Nov 2. PMID 21045179
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between September 2005 and February 2009 in Rochester, Minnesota.
Pre-assignment Details: 969 subjects completed imaging and met eligibility criteria, but 33 were excluded because of lack of the reference standard (unverified cancer status).
Groups:
- Mammography and Molecular Breast Imaging: Participants underwent conventional mammography and molecular breast imaging after a 740-millibecquerel (mBQ)(20-mCi) Technetium (99mTc) sestamibi injection.
Period: Overall Study
Arm/Group | Mammography and Molecular Breast Imaging
Started | 969
Completed | 936
Not Completed | 33
Not completed — Unverified cancer status | 33

BASELINE CHARACTERISTICS:
Groups:
- Mammography and Molecular Breast Imaging: Participants underwent conventional mammography and molecular breast imaging after a 740-mBQ (20-mCi) Technetium (99mTc) sestamibi injection.
Arm/Group | Mammography and Molecular Breast Imaging
Number analyzed (Participants) | 969
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [25 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 969
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 969
Race or ethnicity [Number; unit: participants]
  White | 860
  Hispanic or Latina | 1
  Black or African American | 1
  Asian | 6
  American Indian or Alaskan Native | 1
  Unknown or data missing | 100
Menopausal status [Number; unit: participants]
  Premenopausal | 324
  Perimenopausal | 65
  Postmenopause | 529
  Surgical menopause | 51
Mammographic breast density [Number; unit: participants] — Eligibility was determined by density assessed on a previous mammogram prior to study entry; mammographic density reported refers to density assessed from the study mammogram.
  participants
    Almost entirely fat | 7
    Scattered fibroglandular densities | 129
    Heterogeneously dense | 702
    Extremely dense | 131
Risk factors [Number; unit: participants] — Although participants may have qualified for multiple risk factor categories, they were assigned to only one risk factor category in this table. These risk factors are listed in order of priority. The last two risk factors with respect to first and second-degree relatives with a history of breast cancer refer to subjects who qualified on the basis of family history but did not meet the Gail or Claus model risk threshold levels.
  The Gail risk model focuses on nongenetic risk factors, with limited information on family history. The Claus risk model focuses on genetic risk factors.
  participants
    Known mutation in BRCA1 or BRCA2 gene | 5
    Prior chest, mediastinal, or auxiliary irradiation | 1
    Prior biopsy showing hyperplasia, etc. | 23
    Gail or Claus model lifetime risk ≥ 20% | 165
    Gail model 5 year risk ≥ 2.5% | 297
    Gail model 5 year risk ≥ 1.6% | 238
    1 first-deg relative with history of breast cancer | 82
    2 second-deg relatives history of breast cancer | 85
    personal history of breast cancer | 73

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield
Description: Diagnostic yield is the likelihood that a test or procedure will provide the information needed to establish a diagnosis. In this case, it is the proportion of women with positive results of a screening test and positive results with the reference standard (verified cancer status).
Time Frame: 12 months after mammography and gamma imaging
Population: The analysis population only included participants with a verified cancer status at 12 months after the initial screening (mammography and gamma imaging).
Measure: Number (95% Confidence Interval); unit: cancers per 1000 women screened
Groups:
- Mammography Only: For this reporting arm, the interpretation and analysis was done with mammography only.
- Gamma Imaging: For this reporting arm, the interpretation and analysis was done with gamma imaging only.
- Both Mammography and Gamma Imaging: For this reporting arm, the interpretation and analysis was done with both mammography and gamma images together.
Arm/Group | Mammography Only | Gamma Imaging | Both Mammography and Gamma Imaging
Number analyzed (Participants) | 936 | 936 | 936
cancers per 1000 women screened | 3.2 [1.1 to 9.4] | 9.6 [5.1 to 18.2] | 10.7 [5.8 to 19.6]
Statistical Analysis 1: Comparison: Mammography Only vs Both Mammography and Gamma Imaging; Significant difference p ≤ 0.05; Test type: Superiority or Other; p = .016, t-test, 2 sided
Statistical Analysis 2: Comparison: Mammography Only vs Gamma Imaging; significant difference p ≤ 0.05; Test type: Superiority or Other; p = .07, McNemar

2. Secondary Outcome: Sensitivity
Description: Sensitivity measures the proportion of actual positives which are correctly identified as such.
Time Frame: 12 months after mammography and gamma imaging
Population: as for outcome 1
Measure: Number; unit: number of cancers diagnosed
Arm/Group | Mammography Only | Gamma Imaging | Both Mammography and Gamma Imaging
Number analyzed (Participants) | 11 | 11 | 11
number of cancers diagnosed
  All cancers | 3 [9.7 to 56.6] | 9 [52.3 to 94.9] | 10 [62.3 to 98.4]
  Invasive cancers | 2 [8.2 to 64.1] | 7 [64.6 to 100] | 7 [64.6 to 100]
  Ductal carcinoma in situ (DCIS) | 1 [4.6 to 69.9] | 2 [15.0 to 85.0] | 3 [30.0 to 95.4]
Statistical Analysis 1: Comparison: Mammography Only vs Both Mammography and Gamma Imaging; For all cancers; significant difference p ≤ 0.05; Test type: Superiority or Other; p = .016, McNemar
Statistical Analysis 2: Comparison: Mammography Only vs Gamma Imaging; For all cancers; significant difference p ≤ 0.05; Test type: Superiority or Other; p = .07, McNemar
Statistical Analysis 3: Comparison: Mammography Only vs Both Mammography and Gamma Imaging; For invasive cancers; significant difference p ≤ 0.05; Test type: Superiority or Other; p = .063, McNemar
Statistical Analysis 4: Comparison: Mammography Only vs Gamma Imaging; For invasive cancers; significant difference p ≤ 0.05; Test type: Superiority or Other; p = .063, McNemar
Statistical Analysis 5: Comparison: Mammography Only vs Both Mammography and Gamma Imaging; For ductal carcinoma in situ; significant difference p ≤ 0.05; Test type: Superiority or Other; p = .5, McNemar
Statistical Analysis 6: Comparison: Mammography Only vs Gamma Imaging; For ductal carcinoma in situ; significant difference p ≤ 0.05; Test type: Superiority or Other; p > .99, McNemar

3. Primary Outcome: Number of Participants With Cancer Diagnosis at 12 Months
Time Frame: 12 months after mammography and gamma imaging
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Mammography and Molecular Breast Imaging
Number analyzed (Participants) | 936
participants
  Invasive cancer | 7
  Ductal carcinoma in situ (DCIS) | 4

4. Secondary Outcome: Specificity
Description: Specificity measures the proportion of negatives which are correctly identified as such.
Time Frame: 12 month after mammography and gamma imaging
Population: The analysis population only included participants with a verified cancer status at 12 months after the initial screening (mammography and gamma imaging). The number of participants negative for breast cancer was 936-11 = 925.
Measure: Number; unit: number of true negatives
Arm/Group | Mammography Only | Gamma Imaging | Both Mammography and Gamma Imaging
Number analyzed (Participants) | 925 | 925 | 925
number of true negatives | 840 [88.8 to 92.5] | 861 [91.3 to 94.5] | 788 [82.8 to 87.3]
Statistical Analysis 1: Comparison: Mammography Only vs Both Mammography and Gamma Imaging; significant difference p ≤ 0.05; Test type: Superiority or Other; p < .001, McNemar
Statistical Analysis 2: Comparison: Mammography Only vs Gamma Imaging; significant difference p ≤ 0.05; Test type: Superiority or Other; p = .069, McNemar

5. Secondary Outcome: Recall Rate
Description: Recall rate was defined as the percentage of participants recalled for follow-up studies initiated because of abnormal findings with mammography or gamma imaging.
Time Frame: 12 months after mammography and gamma imaging
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mammography Only | Gamma Imaging | Both Mammography and Gamma Imaging
Number analyzed (Participants) | 936 | 936 | 936
percentage of participants | 9 [7.7 to 11.4] | 8 [6.1 to 9.5] | 15 [13.1 to 17.7]
Statistical Analysis 1: Comparison: Mammography Only vs Both Mammography and Gamma Imaging; significant difference p ≤ 0.05; Test type: Superiority or Other; p < .001, McNemar
Statistical Analysis 2: Comparison: Mammography Only vs Gamma Imaging; significant difference p ≤ 0.05; Test type: Superiority or Other; p = .218, McNemar

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events while they were on the study.
Arm/Group | Mammography and Molecular Breast Imaging
Serious Adverse Events (participants affected / at risk) | 0/969
Other Adverse Events (participants affected / at risk) | 0/969

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No